CLINICAL TRIAL: NCT04257292
Title: NExt-Generation Sequencing and Cell Culture-based Characterization of S. Aureus in Infective Endocarditis
Acronym: NESSIE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Jena University Hospital (Other)
Collaborators: Fraunhofer Institute for Cell Therapy and Immunology, Leipzig, Germany (Unknown)
Responsible Party: Principal Investigator, Mahmoud A. Diab, Dr. med.; Principal Investigator, Jena University Hospital
Other Study IDs: 01
Record Dates: First submitted 2019-09-05; First posted 2020-02-06 (Actual); Last update posted 2020-02-06 (Actual); Status verified 2020-02

CONDITIONS: Infective Endocarditis; Infection Staphylococcal
Keywords: Infective Endocarditis; Staphylococcus aureus; Next-Generation Sequencing
MeSH Terms: conditions — Endocarditis; Staphylococcal Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Isolated strains of S. aureus from blood culture and valve tissue from patients treated for infective endocarditis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Infective endocarditis is a deadly disease with a mortality rate between 20 and 40%. Antibiotic therapy is of utmost importance. It is primarily guided by microbial results from positive blood culture. However, culture-based microbiological diagnostic can identify the species, but not the strain or the genotypic characteristics of a pathogen. Identifying the strain can be of utmost clinical significance. S. aureus is the most common causative organism of IE worldwide (16%-32%). This pathogen causes massive valve destruction and abscesses, which is strongly dependent on the expression of virulence factors that vary between different S. aureus strains.

Functional characterization of S. aureus and determination of virulence factors can currently be achieved through cell culture-based assays (CCBA). However, these tests are very time consuming and cannot be performed as routine clinical diagnostics. Next Generation Sequencing (NSG) has the potential to identify the genotypic characteristics of the pathogen, which is important to determine its virulent potential.

The aim of this study is to evaluate the possible utilization of NGS in the prediction of virulence factors of S. aureus and to compare it to the virulence factors determined using CCBA.

Hopefully, by comparing the NGS and CCBA, the investigators will get a faster way of determining the possible virulence factors. The NGS method can be further utilized to describe the prevalence of different strains of bacteria in infected valve tissue and blood culture samples. The collected data will serve as a basis for further evaluation of the potentials of NGS-based Diagnosis of IE, as well as a comparison between NGS-guided antibiotic treatment and the standard of care antibiotic treatment.

DETAILED DESCRIPTION:
The ability of the Staphylococcus aureus to produce massive valve destruction as well as abscesses and to switch from acute to chronic infection and vice versa is a significant issue in the modern treatment of infective endocarditis. Furthermore, the ability to produce different virulence factors to evade the immune defense mechanisms proves the treatment more difficult. Another conundrum is the proof of different S. aureus strains isolated from Blood culture samples and infected valve samples. This makes a possible treatment of S. aureus-based endocarditis more difficult than expected.

Isolation of Bacteria in the Blood culture samples can take much time (3-14 days), and Cell Culture-based assays (CCBA) are not regularly implemented as a diagnostic procedure. CCBA is not regularly used in the clinical setting due to the time consumption and high cost. The significance of the CCBA method lies in the determination of the possible virulence factors. Utilizing the Next Generation Sequence (NGS) method, it might be possible to gain this information about the culprit microorganism faster and to identify the different strains and virulence factors.

To date, such correlations between genetic information about virulence factors gained by NGS and phenotypic information obtained by cell culture-based assays have not yet been performed.If proven, the NGE based analysis of the pathogens and their phenotypical behavior could guide antimicrobial therapy and make it individualized. Blood culture and infected tissue valve samples will be examined using the NGS and CCBA. The investigators aim to compare the differences in virulence factor results in these two methods, to characterize the prevalence of different strains of S. aureus in the blood culture and valve samples and to evaluate the possible potentials of NGS-based diagnosis of IE and to compare the effects of the NGS-guided antimicrobial therapy to the standard of care therapy.

ELIGIBILITY:
Inclusion Criteria:

* patients with the diagnosis infective endocarditis and indication for heart surgery on a heart valve
* signed informed consent
* age ≥18 years
* pathogens (S. aureus) can be isolated from blood culture AND from the removed valve tissue

Exclusion Criteria:

* S. aureus can not be isolated from removed valve tissue

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with the diagnosis infective endocarditis and indication for heart surgery on a heart valve
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-02-28 (Estimated); Study Completion 2020-07-31 (Estimated)

PRIMARY OUTCOMES:
biofilm growth | through study completion (about 1 year)
  ability of S. aureus strains isolated from the blood and heart tissue of included patients to build a biofilm

SECONDARY OUTCOMES:
invasion characteristics | through study completion (about 1 year)
  characteristics of the S. aureus strains isolated from the blood and heart tissue of included patients to invade other cells (host cell invasion; persistence in host cells; tests will be conducted in cell culture)
adhesion characteristics | through study completion (about 1 year)
  characteristics of the S. aureus strains isolated from the blood and heart tissue of included patients to adhere to other human cells (important information regarding the ability to attach to heart tissue; test will be conducted in cell culture)
toxine production | through study completion (about 1 year)
  characteristics of the S. aureus strains isolated from the blood and heart tissue of included patients regarding production of toxins which will lead to information about induction of inflammation processes and induction of host cell death

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud A Diab, Dr. med., Principal Investigator — Jena University Hospital, Clinic for Cardiac and Thoracic Surgery
Locations (1):
- Jena University Hospital, Clinic for Cardiothoracic surgery, Jena, Germany

IPD SHARING:
Plan to Share IPD: Undecided